CLINICAL TRIAL: NCT06638658
Title: Postoperative Complications of Orthopedic Surgery in Patients From High-altitude Regions: a Cohort Study.
Brief Title: Postoperative Complications of Orthopedic Surgery in Patients From High-altitude Regions
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: 20241284
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Orthopedic Surgery; Postoperative Complications; High Altitude
Keywords: High-altitude population; Perioperative cohort; Orthopedic surgery
MeSH Terms: conditions — Postoperative Complications; Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and hair.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic surgery patients from high-altitude regions: high altitude patients Undergoing orthopedic surgery

SUMMARY:
This study will focus on orthopedic surgery patients from high-altitude regions, utilizing smart wearables and monitoring tools to gather perioperative data, including heart rate, oxygen saturation, sleep quality, stress levels, and other relevant metrics. Regular follow-ups will assess recovery and complications, in addition to collecting medical records, lab results, imaging data, and other pertinent records. The ultimate goal is to establish a comprehensive follow-up cohort of orthopedic surgery patients from high-altitude areas.

DETAILED DESCRIPTION:
Prolonged exposure to hypoxic and low-pressure environments leads to structural remodeling and functional abnormalities in the cardiovascular, respiratory, and hematological systems of high-altitude populations. This elevates the risk of postoperative complications, particularly in patients undergoing orthopedic surgery, significantly impacting their recovery and quality of life. This study will focus on orthopedic surgery patients from high-altitude regions. Using smart wearable devices and other monitoring tools, comprehensive perioperative dynamic data of participants, including heart rate, heart rate variability, oxygen saturation, respiratory rate, sleep quality, activity levels, stress index, and other relevant indicators will be collected. Regular follow-ups will be conducted to evaluate postoperative recovery and monitor the incidence of perioperative complications. Additionally, perioperative data such as electronic medical records, laboratory test results, ECG waveforms, echocardiography, chest CT images, and other pertinent records will be also collected. Through that, this study aims to establish a follow-up cohort of orthopedic surgery patients from high-altitude regions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. ASA classification I-III;
3. Patients who have lived at an altitude above 2500 meters for more than 6 months ;
4. Patients scheduled for elective orthopedic surgery.

Exclusion Criteria:

1. Urgent or emergent surgery;
2. Expected hospital stay < 48 hours;
3. Inability to provide informed consent；
4. Patients who have been out of high-altitude regions for over three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have lived in high-altitude regions scheduled for orthopedic surgery.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative venous thromboembolism | During hospitalization
  Defined according to the European Perioperative Clinical Outcome (EPCO) criteria, including both deep vein thrombosis and pulmonary embolism.

SECONDARY OUTCOMES:
Postoperative venous thromboembolism | Up to 2 weeks postoperatively
  Defined according to the European Perioperative Clinical Outcome (EPCO) criteria, including both deep vein thrombosis and pulmonary embolism.
A composite of postoperative pulmonary complications | During hospitalization
  Defined according to the European Perioperative Clinical Outcome (EPCO) criteria, including respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonia.
Postoperative major adverse cardiovascular events | During hospitalization
  Defined according to the European Perioperative Clinical Outcome (EPCO) criteria, including non-fatal cardiac arrest, acute myocardial infarction, congestive heart failure, new cardiac arrhythmias, angina, et al.
Postoperative nausea and vomiting | During hospitalization
  Nausea and vomiting
The quality of postoperative recovery | During hospitalization
  Assessed using QoR-15 score at different time points after surgery
Chronic pain after surgery | Up to 1 year postoperatively
  Assessed using NRS scale and BPI at different time points after surgery
Postoperative quality of life assessment | Up to 1 year postoperatively
  Assessed using WHODAS2.0 scores at different time points after surgery

OTHER OUTCOMES:
Pain scores of movement-evoked pain | During hospitalization
  Assessed using NRS scale and BPI at different time points after surgery
Pain scores at rest | During hospitalization
  Using NRS scale and BPI at different time points after surgery
Surgical site infection | During hospitalization
  Defined according to the European Perioperative Clinical Outcome (EPCO) criteria
Time of Bowel function recovery | During hospitalization
  Defined as time to first defecation or flatus
Sleep quality after surgery | Up to 1 year postoperatively
  Assessed using the Pittsburgh Sleep Quality Index (PSQI) and the Morningness-Eveningness Questionnaire (MEQ) at different time points after surgery
Postoperative anxiety assessment | Up to 1 year postoperatively
  Assessed using GAD-7 scores at different time points after surgery
Postoperative depression assessment | Up to 1 year postoperatively
  Assessed using PHQ-9 scores at different time points after surgery
Postoperative cognitive function assessment | Up to 1 year postoperatively
  Assessed using AD-8 and three-word recall test scores at different time points after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: Undecided